CLINICAL TRIAL: NCT04984759
Title: Breastfed Child Exposure to Tafenoquine and Primaquine During Treatment in Lactating Women: a Pharmacokinetic Study in Healthy Volunteers
Brief Title: Tafenoquine and Primaquine in Colostrum and Breast Milk
Acronym: TBM
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Local EC requested that the arms of study be submitted as separate protocols so they could respond to the different risk of each arm. In response investigators have withdrawn this protocol and begun separate submissions, starting with NCT06191458.
Sponsor: University of Oxford (Other)
Collaborators: Mahidol Oxford Tropical Medicine Research Unit (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MAL21004
Record Dates: First submitted 2021-07-14; First posted 2021-08-02 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-03

CONDITIONS: Healthy Lactating Women
Keywords: Healthy lactating women; Tafenoquine; Primaquine; Plasmodium Vivax; Pharmacokinetic
MeSH Terms: conditions — Malaria, Vivax | interventions — Primaquine; tafenoquine

STUDY DESIGN:
Intervention Model Description: Arms 1 and 2 will enroll first as preliminary data from Arms 1 and 2 is needed before Arm 3 can begin enrolment.
  All eligible and consenting women who are immediately postpartum will be enrolled in Arm 1 until it is completed.
  Arm 2 will enroll eligible women breastfeeding older infants and young children. If there are no safety concerns after 2-4 mother-child dyads have been enrolled in Arm 2, successively younger infants will be enrolled to a minimum of 14 days old.
  If there are no safety concerns with Arms 1 and 2, Arm 3 will begin enrolment.
Masking Description: This is a prospective open-label study in which both participants and investigators know the identity of the treatment and its dosage.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Primaquine in colostrum and transitional milk (mother-neonate pairs) (Experimental): 12 women who are breast feeding neonates ≤5 days old will be recruited into the primaquine arm. They will receive primaquine 0.5 mg/kg daily for 14 days directly observed in the clinic.
  Interventions: Drug: Primaquine
- Tafenoquine in mature milk (mother-child pairs) (Experimental): 24 women who are breast feeding infants or young children > 14 days will be recruited into Arm 2. They will receive a single 300 mg dose of tafenoquine directly observed in the clinic. Investigators will begin with recruiting 2-4 women breastfeeding young children ≥12 months old.
  Interventions: Drug: Tafenoquine
- Tafenoquine in colostrum and transitional milk (mother-neonate pairs) (Experimental): 12 women who are breast feeding neonates ≤ 5 days old will be recruited into Arm 3. They will receive a single 300 mg dose of tafenoquine directly observed in the clinic.
  Interventions: Drug: Tafenoquine

INTERVENTIONS:
Drug: Primaquine — Primaquine GPO® (Government Pharmaceutical Organization (GPO), Thailand) 0.5 mg/kg will be given once daily with food for 14 days. This is the dose recommended for radical cure of P. vivax in tropical areas with high rates of relapse, such as the study design setting. Doses will be directly supervised (DOT).
  Other Names: Primaquine GPO®
  Arms: Primaquine in colostrum and transitional milk (mother-neonate pairs)
Drug: Tafenoquine — Tafenoquine (Kodatef, Biocelect Pty Ltd.) 300 mg will be given as a directly observed single dose with food. This is the standard dose recommended globally for radical cure of P. vivax.
  Other Names: Kodatef
  Arms: Tafenoquine in colostrum and transitional milk (mother-neonate pairs); Tafenoquine in mature milk (mother-child pairs)

SUMMARY:
Each year almost a million infants are born small for gestational age due to malaria infection in pregnancy. These infants are at risk for stillbirth or neonatal death, and being born too small predisposes the survivors to increased metabolic diseases later in life. Plasmodium vivax (PV) is the second most common malaria species globally. Its relapsing nature results in multiple episodes of PV in a single pregnancy, compounding growth restriction and stillbirth risk. Women with PV in one pregnancy may harbor dormant parasites (hypnozoites) in their liver the cause illness and poor fetal growth in a subsequent pregnancy.

Only radical cure with 8-aminoquinolines (8AQ)- primaquine (PMQ) or tafenoquine (TQ) - can eliminate hypnozoites, but these drugs are contraindicated in pregnancy. The postpartum period presents a key window of opportunity for giving radical cure to women of childbearing age with PV. Pharmacokinetic data is needed to support safe use of these drugs postpartum and World Health Organization has identified pharmacokinetic studies of 8AQ in lactation as a research priority.

Primaquine is excreted minimally in mature breast milk, at <1% of the weight-adjusted relative infant dose (RID). As the main adverse event associated with both 8AQ - hemolysis glucose-6-phosphate dehydrogenase (G6PD) deficient individuals - is dose-dependent and negligible at low doses, this finding strongly supports its safe use in later lactation. This study is needed to determine if primaquine can also be given safely in the early postpartum period. There is no published data on tafenoquine excretion in breastmilk, and this study would quantify safety throughout early and late lactation.

Drug safety studies in lactation are essential to ensure medications are not denied and unnecessary interruption of breastfeeding is avoided. Demonstration of safety of radical cure for breastfeeding women in the postpartum period would allow women with PV in pregnancy and lactation to receive 8AQ after delivery, preventing illnesses in the postpartum period and subsequent pregnancies. Improved uptake of radical cure through elimination of unnecessary contraindications supports malaria elimination and community health.

The main purpose of this study is to characterize the transfer of tafenoquine and primaquine in breast milk of mothers receiving radical cure doses of 8AQ throughout the different phases of lactation - colostrum, transitional milk, and mature milk - in order to determine the degree of infant exposure.

DETAILED DESCRIPTION:
The study will take place at clinics of the Shoklo Malaria Research Unit (SMRU), Mahidol-Oxford Tropical Medicine Research Unit in Tak Province, Thailand. The clinics serve a population of migrant workers resident along the Thailand-Myanmar border. Non-pregnant breastfeeding women that access care at SMRU (postnatal care, outpatient, vaccine and routine baby care departments) will be invited to participate with their breastfed children.

All lactating women and their children will be G6PD phenotypically normal. Participants will be enrolled as follows; Arm 1: Primaquine mother-neonate pairs Arm 2: Tafenoquine mother-child pairs Arm 3: Tafenoquine mother-neonate pairs

Pharmacokinetic sampling plan:

* PMQ pharmacokinetic sampling (Mother/Neonate pairs - Arm 1):

  * Mothers: Dense pharmacokinetic venous blood and breast milk sampling will be performed during day 1 and 14; one sample of blood and breast milk will collected at a single timepoint on days 3, 5 and 8.
  * Neonate: One capillary blood sample will be collected on the same days as maternal sampling.
* TQ pharmacokinetic sampling (Mother/child pairs - Arms 2, and 3):

  * Mothers: Dense pharmacokinetic venous blood and breast milk sampling will be performed during the first day after dosing, followed by one sample of blood and breast milk at a single time point on days 2, 3, 8, 15, 29, 43 and 75 (allowing a description of approximately 95% of the total drug exposure).
  * Child: One capillary blood sample will be collected on the same days as maternal sampling.

Mothers and children will be closely monitored for safety throughout the 75 day follow up period including regular assessments of adverse events, Hb, Hct and MetHb levels. Pharmacokinetic drug measurements of primaquine, carboxyprimaquine and tafenoquine will be performed at the Department of Clinical Pharmacology, Mahidol-Oxford Tropical Medicine Research Unit (MORU), Bangkok, Thailand. Drug concentrations will be quantified by liquid chromatography coupled with tandem mass spectrometry (LC-MS/MS). Interim data review will be done by an external drug safety monitoring board (DSMB) before recruitment of Arm 3. The board will review safety data and any available PK data. If PK data is not yet available and there are safety concerns, recruitment in Arm 3 may be suspended until PK data from Arms 1 and 2 are available.

Study participants with any adverse events will be followed until the event has stabilized or resolved (unless the participant refuses such follow up care). Free care will be offered through SMRU clinics. For severe harm caused by study procedures following this protocol, Oxford University insurance will support additional health care beyond SMRU's capacity.

This study is funded by Thrasher Research Fund.

ELIGIBILITY:
Inclusion Criteria:

* Mother

  * Lactating women >= 16 years old who are breast feeding one child who fits the time window for the respective study arm
  * Planning to breastfeed for the duration of the study
  * Willingness and ability to comply with the study protocol for the duration of the study
  * Willingness to delay pregnancy until the end of the period of drug exposure (14 days for PMQ and 90 days for TQ)
  * Current pregnancy excluded by urine pregnancy test and ultrasound OR immediate postpartum status (≤2 months)
  * Can understand information about the study and provide consent
* Children

  * Healthy children falling into the time window for the respective study arm
  * ≤ 5 days for Arms 1 & 3
  * > 14 days for Arm 2

Exclusion Criteria:

* Mothers

  * Known hypersensitivity to PMQ or TQ, defined as history of erythroderma/other severe cutaneous reaction, angioedema or anaphylaxis
  * Known Glucose-6-phosphate-dehydrogenase (G6PD) deficiency in mother defined as G6PD activity <70% of normal male population median by spectrophotometry
  * Presence of any condition which in the judgement of the investigator would place the participant at undue risk or interfere with the results of the study
  * Alkaline phosphatase (ALT) > 2x the upper limit of normal (ULN)
  * Pregnancy
  * Screening hematocrit (Hct) <33%
  * Known history of severe jaundice in a previous child
  * Known history of psychiatric illness or abnormal depression screening score
  * Blood transfusion within the 3 months before screening
* Children

  * Known hypersensitivity to primaquine or tafenoquine, defined as history of erythroderma/other severe cutaneous reaction, angioedema or anaphylaxis
  * Known Glucose-6-phosphate-dehydrogenase (G6PD) deficiency in child defined as G6PD activity <70% of normal male population median by spectrophotometry in children
  * Presence of any condition which in the judgement of the investigator would place the participant at undue risk or interfere with the results of the study
  * Screening Hct <33%
  * Estimated gestational age at birth < 38 weeks
  * Blood transfusion within the 3 months before screening
  * Evidence of birth asphyxia (5 min Apgar score <7)
  * Moderate or severe jaundice as defined as total serum bilirubin above treatment line on day 1 (before maternal dose)

Min Age: 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Lactating women >= 16 years old who are breast feeding one child who fits the time window for the respective study arm
Enrollment: 0 (Actual)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
To characterize the excretion of tafenoquine and primaquine (with its main metabolite, carboxyprimaquine) in colostrum, transitional milk and mature milk in order to determine the degree of infant exposure | Days 1-14 for primaquine, Days 1-75 for tafenoquine
  End points: Area under the time-concentration curve (AUC) for 8-aminoquinolines in colostrum, transitional milk and mature milk.
  Relative infant dose (RID) for 8-aminoquinolines calculated using AUCs for drug in maternal plasma and colostrum, transitional milk and mature milk.

SECONDARY OUTCOMES:
To evaluate the pharmacokinetics (PK) of primaquine and tafenoquine in lactating women and their breastfed children at different time points following delivery. | Days 1-14 for primaquine, Days 1-75 for tafenoquine
  End point: AUC of tafenoquine and primaquine for mother and child (if measurable concentrations found in child plasma).
To evaluate the pharmacokinetics (PK) of primaquine and tafenoquine in lactating women and their breastfed children at different time points following delivery. | Days 1-14 for primaquine, Days 1-75 for tafenoquine
  End point: Time to maximum concentration (Tmax) of tafenoquine and primaquine for mother and child (if measurable concentrations found in child plasma).
To evaluate the pharmacokinetics (PK) of primaquine and tafenoquine in lactating women and their breastfed children at different time points following delivery. | Days 1-14 for primaquine, Days 1-75 for tafenoquine
  End point: Maximum concentration reached (Cmax) of tafenoquine and primaquine for mother and child (if measurable concentrations found in child plasma).
To describe hematologic changes in mothers and breastfeed children during maternal ingestion of radical cure doses of 8-aminoquinolines. | Days 1-75
  End points: Changes in hemoglobin (Hb), hematocrit (Hct) and methemoglobin (MetHb) in mothers and children over the period of drug exposure.
To assess adverse events of maternal radical cure doses of 8-aminoquinolines in mothers and their breastfeeding children. | Days 1-75
  End points: Number, severity and type of adverse events in mothers and children during the period of drug exposure.

CONTACTS AND LOCATIONS:
Overall Officials: Rose McGready, Ph.D, Principal Investigator — Shoklo Malaria Research Unit (SMRU), PO Box 46, 68/30 Ban Toong Road, Mae Sot, Tak 63110
Locations (1):
- Shoklo Malaria Research Unit (SMRU), Mae Sot, Changwat Tak, Thailand

IPD SHARING:
Plan to Share IPD: Yes
All data will be published in the open access medical literature with the identity of the participants protected. Criteria for authorship will follow international guidelines. Following completion of the study, the database will belong to the PI and key co-investigators. The database, including individual participant data, may be shared with researchers not directly involved with the study after the original research has been published and in accordance with SMRU and MORU data sharing policies. The results of the study will be shared with the local community.
Time Frame: After completion of the study
Access Criteria: SMRU and MORU Data Sharing Policies
  The criteria for authorship will be consistent with the international guidelines (http://www.icmje.org/#author).
URL: https://www.tropmedres.ac/units/moru-bangkok/bioethics-engagement/data-sharing